CLINICAL TRIAL: NCT02451475
Title: Comparative Effectiveness of Newer Antidepressants in Combination With Pregabalin for Fibromyalgia Syndrome: A Controlled Randomized Study
Brief Title: Newer Antidepressants in Combination With Pregabalin for Fibromyalgia Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed R El Tahan, Associate Professor, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MUH-ANES-2013-10
Record Dates: First submitted 2015-05-16; First posted 2015-05-22 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Fibromyalgia
Keywords: Pregabalin; Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Amitriptyline; Venlafaxine Hydrochloride; Paroxetine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Amitriptyline (Other): Amitriptyline 25 mg/day
  Interventions: Drug: Amitriptyline
- Venlafaxine (Active Comparator): Venlafaxine 75 mg/day
  Interventions: Drug: Venlafaxine
- Paroxetine (Active Comparator): Paroxetine 25 mg/day
  Interventions: Drug: Paroxetine

INTERVENTIONS:
Drug: Amitriptyline — Amitriptyline 25 mg/day
  Arms: Amitriptyline
Drug: Venlafaxine — Venlafaxine 75 mg/day
  Arms: Venlafaxine
Drug: Paroxetine — Paroxetine 25 mg/day
  Arms: Paroxetine

SUMMARY:
Background: The investigator hypothesized that the combined use of pregabalin and paroxetine would be associated with comparable Somatic Symptoms Scale-8 (SSS-8) and higher tolerability than amitriptyline or venlafaxine.

Methods: After ethical approval, 75 patients with diagnosed fibromyalgia who were receiving pregabalin 75 mg/day, were randomly allocated to receive amitriptyline 25 mg/day (n = 24), venlafaxine 75 mg/day (n = 25), or paroxetine 25 mg/day (n = 26). All patients were assessed bi-monthly for consequent six months for the changes in the SSS-8, Center for Epidemiological Studies Depression Scale (CESDS), life satisfaction, mood, sleep quality, fatigue and medication tolerability and adverse effects.

DETAILED DESCRIPTION:
Fibromyalgia is a common cause of chronic widespread disabling pain affecting 2-5% of the young to middle-aged women in developed countries. The American College of Rheumatology has been established new diagnostic criteria for fibromyalgia in 2010 included a widespread pain index (WPI) and categorical scales for cognitive symptoms, unrefreshed sleep, fatigue, and number of somatic symptoms. The definite pathophysiology of chronic pain in fibromyalgia remains unclear.

Fibromyalgia is usually associated with depression, anxiety, and alexithymia increasing over age which contribute significantly to reduced patient wellbeing. These may be due to alterations of central pain pathways, hyporeactivity of the hypothalamus-pituitary-adrenal axis, and disturbances in the dopaminergic and serotonergic systems. Thus the European League Against Rheumatism (EULAR) recommends the use of serotonin and noradrenaline reuptake inhibitors (SNRIs) for the treatment of fibromyalgia, to reduce pain and improve function.

However, few patients achieve satisfactory pain relief with the sole use of SNRIs. A recent Cochrane review demonstrated only modest improvement in relieving pain without reducing of sleep disturbances, fatigue, or the poor quality of life with the use of duloxetine and milnacipran than placebo in patients with fibromyalgia. More patients experienced adverse events like as nausea, dry mouth, constipation, headache, somnolence, dizziness and insomnia leading to stopping medications. Whereas, the evidence from clinical studies shows that combined use of pregabalin and SNRIs such as duloxetine has potential efficacy and better tolerability during the treatment of improvement of pain, fatigue, and sleep disorders in patients with fibromyalgia.

The use of the second-generation antidepressants like as paroxetine (a selective serotonin reuptake inhibitors (SSRIs)) and venlafaxine (SNRIs) may be associated with more tolerability and reduce pain in patients with major depressive disorder.

To the best of the investigator's knowledge, the comparison of the long-term efficacy, tolerability, and safety of the combined use of pregabalin with one of the three antidepressants, namely, amitriptyline, venlafaxine, or paroxetine for the treatment of fibromyalgia has not yet been studied.

The investigators hypothesized that the combined use of pregabalin and paroxetine would be associated with comparable Somatic Symptoms Scale-8 (SSS-8) and Center for Epidemiological Studies Depression scales (CESD) and higher tolerability than the use of pregabalin with either amitriptyline or venlafaxine.

ELIGIBILITY:
Inclusion Criteria:

* Fibromyalgia
* Receiving pregabalin daily

Exclusion Criteria:

* Pathologies mimicking the symptoms of fibromyalgia
* Acute systemic inflammatory diseases
* Infections
* Pregnancy
* Lactating

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2013-02; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Somatic Symptoms Scale-8 (SSS-8) | for six months after start of the medication
  Using the 8-points Somatic Symptoms Score

SECONDARY OUTCOMES:
Center for Epidemiological Studies Depression (CSED) | for six months after start of the medication
  According to the Center for Epidemiological Studies Depression (CSED) questionnaire
Life satisfaction | for six months after start of the medication
  Using a life satisfaction score
Mood | for six months after start of the medication
  Using a mood score
Sleep quality | for six months after start of the medication
  Using a sleep quality questionnaire
Fatigue | for six months after start of the medication
  Using a fatigue questionnaire
Tolerability | for six months after start of the medication
  Using a tolerability questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Eiad Ramzy, MD, Principal Investigator — Lecturer of Anesthesia and Surgical ICU, Mansoura University , Mansoura City, Egypt